CLINICAL TRIAL: NCT00776698
Title: An Open Label Study to Establish the Preferred Dose and to Assess Safety and Overall Response Rate of Avastin in Combination With Concomitant Thoracic Radiation and Chemotherapy (Cisplatin and Etoposide) in Locally Advanced Unresectable Non-squamous Non-small Cell Lung Cancer.
Brief Title: A Study of Avastin (Bevacizumab) in Combination With Thoracic Radiation and Chemotherapy in Patients With Advanced Non-Squamous Non-Small Cell Lung Cancer.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BO21563; 2008-002279-28
Record Dates: First submitted 2008-10-20; First posted 2008-10-21 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — Bevacizumab; Cisplatin; Etoposide

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: bevacizumab [Avastin]; Drug: cisplatin; Drug: etoposide

INTERVENTIONS:
Drug: bevacizumab [Avastin] — 7.5mg/kg every 3 weeks for 3 cycles (cohort 1) or 15mg/kg every 3 weeks for 3 cycles (cohort 2). Preferred dose every 3 weeks for 9 cycles (cohort 3).
Drug: cisplatin — 80mg/m2 iv every 3 weeks for 3 cycles
Drug: etoposide — 100mg/m2 iv for 3 consecutive days, every 3 weeks for 3 cycles

SUMMARY:
This single arm study will evaluate the feasibility of treatment with 2 dose levels of Avastin in combination with concurrent thoracic radiation and chemotherapy in patients with locally advanced unresectable non-squamous non-small cell lung cancer. Two cohorts of patients will receive 3 cycles of Avastin treatment (7.5mg/kg and 15mg/kg iv every 3 weeks, respectively), concurrently with thoracic radiation and chemotherapy (cisplatin and etoposide). Once a preferred dose has been established, this dose will be applied to a 3rd cohort, who will then receive maintenance treatment with Avastin as a single agent for 6 additional cycles. The anticipated time on study treatment is <3 months for cohorts 1 and 2, and 3-12 months for cohort 3, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >= 18 years of age;
* non-squamous non-small cell lung cancer, locally advanced and unresectable;
* ECOG performance status 0 or 1;
* no prior thoracic or head and neck radiation;
* no prior surgical resection for current lung cancer.

Exclusion Criteria:

* malignancies other than non-small cell lung cancer within 2 years prior to inclusion, except for basal cell cancer of the skin, squamous cancer of the skin, or cancer in situ of the cervix;
* prior systemic therapy for non-small cell lung cancer;
* clinically significant cardiovascular disease;
* history of >= grade 2 hemoptysis;
* current or recent use of aspirin (>325mg/day) or full dose anticoagulants or thrombolytic agents for therapeutic purposes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2009-04; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity | Throughout Study

SECONDARY OUTCOMES:
AEs, laboratory parameters | Throughout Study
Tumor response | Throughout Study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- Netherlands (3):
  - Amsterdam
  - Groningen
  - Maastricht
- United Kingdom (2):
  - Aberdeen
  - Manchester